CLINICAL TRIAL: NCT04500015
Title: Benefits of Self-administered Vaginal Isonicotinic Acid Hydrazide (INH) Administration 12 Hours Prior to Intrauterine Device Insertion in Adolescent and Young Women: a Randomized Controlled Trial
Brief Title: Vaginal Isonicotinic Acid Hydrazide Administration Prior to Intrauterine Device Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/354/4/19
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: IUCD Complication

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 vaginal tablet of isonicotinic acid hydrazide self-inserted by the patient 12 hours before IUD insertion.
  Interventions: Drug: INH
- Placebo Comparator (Placebo Comparator): 3 tablet of placebo self-administered by the patient 12 hours before IUD insertion
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: INH — 3 vaginal tablet of isonicotinic acid hydrazide self-inserted by the patient 12 hours before IUD insertion.
  Arms: INH
Drug: Placebo Comparator — 3 tablet of placebo self-inserted by the patient 12 hours before IUD insertion.
  Arms: Placebo Comparator

SUMMARY:
To investigate whether vaginal isonicotinic acid hydrazide administered before the levonorgestrel-releasing intrauterine system insertion reduces IUD insertion pain and difficulty in insertion in adolescents and young women.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous adolescent and young women requesting levonorgestrel-releasing intrauterine device

Exclusion Criteria:

* pregnancy and
* contraindication or allergy to or contraindication to IUD insertion,
* chronic pelvic pain,
* pelvic inflammatory disease,
* analgesic intake 24 hours prior to IUD insertion.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — adolescents and young women.
Enrollment: 130 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

SECONDARY OUTCOMES:
duration of IUD insertion | 10 minutes
  duration of IUD insertion measured in minutes
Provider ease of insertion | 10 minutes
  Provider ease of insertion was evaluated using a visual analog scale from 0 to 10 cm where 0 denotes very easy insertion and 10 denotes a very difficult insertion.

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No